CLINICAL TRIAL: NCT06041334
Title: Evaluation of muLtimodal and Non-invasive SPINa Bifida Neurovessels During Prospective Follow-up
Acronym: SPINLESS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Collaborators: NeuroSphinx (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 35RC20_9746_SPINLESS; IDRCB (Other: 2022-A02780-43)
Record Dates: First submitted 2023-09-07; First posted 2023-09-18 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Spina Bifida
Keywords: Spina Bifida; urinary biomarker; upper urinary tract; Galloway score; urodynamic work-up; urethrocystography
MeSH Terms: conditions — Spinal Dysraphism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study volunteers (Other)
  Interventions: Biological: Collection of a urine sample; Diagnostic Test: Magnetic Resonance Imaging of the bladder

INTERVENTIONS:
Biological: Collection of a urine sample — Collection of a urine sample for analysis of urinary biomarkers and urinary metabolomics (Inclusion and 1 year)
Diagnostic Test: Magnetic Resonance Imaging of the bladder — Magnetic Resonance Imaging of the bladder (10 adults patients only) (Inclusion and 1 year)

SUMMARY:
The aim of the study is to investigate known urinary biomarkers in order to determine whether they can be predictive of a risk of damage to the upper urinary tract and therefore the kidneys in patients with spina bifida. The risk of damage to the upper urinary tract can be calculated using the Galloway score, based on the results of the urodynamic study and retrograde urethrocystography, which all patients with spina bifida have regularly.

The urinary biomarkers studied TIMP-2 (Tissue inhibitor of metalloproteinases 2) and MMP-2 (matrix metalloproteinase-2) are potentially associated with renal degradation, but this has not yet been demonstrated.

Volunteers to take part in the study will have their biomarkers measured at the time of their urodynamic assessment.

ELIGIBILITY:
Inclusion Criteria:

* Spina patients consulted as part of the multidisciplinary consultation of the spina bifida rare disease reference centre;
* Written consent to participate in the research.
* Compulsory membership of a social security scheme

Exclusion Criteria:

* Patients with a non-continuous trans ileal urinary diversion ;
* Patients with enterocystoplasty;
* Untreated bacteriuria at the time of urodynamic assessment and urine sample collection;
* History of urinary tract tumour;
* History of histologically proven interstitial cystitis;
* Persons under legal protection (safeguard of justice, curatorship, guardianship);
* Persons deprived of their liberty.
* Women claiming to be pregnant

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-01-18 (Actual); Primary Completion 2027-07-18 (Estimated); Study Completion 2028-07-18 (Estimated)

PRIMARY OUTCOMES:
Verify if levels of urinary biomarkers Metalloproteinase Inhibitor 2 and matrix metalloproteinase-2 are associated with Galloway score | 1 day
  Logistic regression based on composite analysis of Galloway score (≤ 5 (low risk) or >5 (high risk)) and the rate of urinary biomarkers.

SECONDARY OUTCOMES:
Galloway score | 1 year
  Change in Galloway score from baseline to 1 year based on change in urinary biomarkers Metalloproteinase Inhibitor 2 and matrix metalloproteinase-2
Success or failure of treatment | 1 year
  The success of the treatment will be assessed at 1 year after its implementation according to an hybrid criteria : In the event of a Patients Global Impression of Improvement for Incontinence questionnaire < 3 and/or a Galloway score reduction of 1 or 2, the treatment will be considered successful.
Relationship between the success of the treatment implemented at inclusion and the level of urinary biomarkers | 1 year
  The relationship between the success of the treatment implemented at inclusion and the level of the urinary biomarkers Metalloproteinase Inhibitor 2 Anticorps and matrix metalloproteinase-2 at inclusion will be studied.
Bladder hypocompliance based on metabolomic profile at inclusion | 0 day
  Presence or absence of bladder hypocompliance on urodynamic assessment at baseline, based on metabolomic profile at baseline.
Bladder hypocompliance based on MRI radiomic markers at inclusion | 0 day
  Presence or absence of bladder hypocompliance on the urodynamic work-up at inclusion, based on MRI radiomic markers at inclusion.
Bladder hypocompliance based on MRI radiomic markers at 1 year | 1 year
  Presence or absence of bladder hypocompliance on urodynamic assessment at 1 year according to MRI radiomic markers at 1 year
Presence of biomarkers on bladder histological specimens | From enrollment to 1 year
  Presence of Metalloproteinase Inhibitor 2 Anticorps and matrix metalloproteinase-2 biomarkers on bladder histological specimens based on levels of urinary Metalloproteinase Inhibitor 2 Anticorps and matrix metalloproteinase-2 biomarkers respectively.

CONTACTS AND LOCATIONS:
Locations (1):
- Rennes University Hospital, Rennes, CHU de Rennes, France

IPD SHARING:
Plan to Share IPD: Undecided